CLINICAL TRIAL: NCT04816305
Title: Project NEUROMOD: Non-invasive Neuromodulation Guided Through Biomarkers in Patients With Stroke Sequels
Brief Title: Non-invasive Neuromodulation Guided Through Biomarkers in Patients With Stroke Sequels
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade Federal de Pernambuco (Other)
Responsible Party: Principal Investigator, Kátia Monte-Silva, Clinical professor, Universidade Federal de Pernambuco
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TMS_biomarkers_stroke
Record Dates: First submitted 2020-10-22; First posted 2021-03-25 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Stroke
Keywords: Transcranial magnetic stimulation; Electroencephalogram; Physiotherapy; Brain symmetry; Biomarker
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- rTMSc + physiotherapy (Experimental): A conventional high-frequency rTMS (rTMSc) will be applied over the lesioned hemisphere over the motor cortex. After rTMSc, patients will be submitted to 45 minutes of neurofunctional physiotherapy. Experimental sessions will be repeated five times per week for two weeks.
  Interventions: Device: rTMSc; Behavioral: Neurofunctional physiotherapy
- rTMSp + physiotherapy (Experimental): A personalized high or low-frequency rTMS (rTMSp) will be applied to the lesioned or non-lesioned hemisphere depending on cortical biomarkers assessment guide a personalized stimulation for each patient in this group. After rTMSp, patients will be submitted to 45 minutes of neurofunctional physiotherapy. Experimental sessions will be repeated five times per week for two weeks.
  Interventions: Device: rTMSc; Behavioral: Neurofunctional physiotherapy
- tDCS sham + physiotherapy (Sham Comparator): The sham protocol will be delivered to each patient of this arm imitating the exat sound of the equipment and structure of the experimental arms. After rTMS sham, patients will be submitted to 45 minutes of neurofunctional physiotherapy. Experimental sessions will be repeated five times per week for two weeks.
  Interventions: Behavioral: Neurofunctional physiotherapy; Device: rTMS sham

INTERVENTIONS:
Device: rTMSc — In all rTMS protocols the patient will remain seated in a comfortable chair with adjustable arms and head rests. Before the start of the conventional rTMS (rTMSc), the resting motor threshold (RMT) of the first dorsal interosseous muscle contralateral to the lesioned hemisphere will be determined. The RMT will be defined as the lowest RMT intensity necessary to produce a motor evoked potential amplitude greater than or equal to 50 µV in at least 5 out of 10 attempts.
  Arms: rTMSc + physiotherapy; rTMSp + physiotherapy
Behavioral: Neurofunctional physiotherapy — All patients will be submitted to a protocol of exercise with different levels according to motor learning, neuroplasticity principles and motor impairment. All physiotherapists will be trained prior to the study.
Device: rTMS sham — During the rTMS sham sessions the same procedures will be used as the rTMSc protocols, however, the magnetic stimulator and its coil will be turned off.
  Arms: tDCS sham + physiotherapy

SUMMARY:
This study aims to investigate if the size effect of repetitive magnetic transcranial stimulation in the paretic upper limb in patients after stroke is influenced by the therapeutic decision.

DETAILED DESCRIPTION:
After the patients and volunteers signed an informed consent form they will be classified and randomized using a website (randomization.com) by a non-involved researcher.

All patients and volunteers will be assigned to groups (arms) after being tried:

(i) rTMS-DIR: in which the patients will be submitted to a customized treatment with repetitive transcranial magnetic stimulation (rTMS) based in neurophysiological assessments; (ii) rTMS: patients will be submitted to standard treatment in the lesioned or non-lesioned hemisphere based in neurophysiological assessments; (iii) rTMS sham: each patient will receive a sham intervention that emits the same sound as the real stimulation;

In each group, the patients will be submitted to 10 sessions for two weeks, five days a week in which will receive the rTMS followed by 45 minutes of neurofunctional physiotherapy. All outcomes will be assessed before and after the 10 sessions.

ELIGIBILITY:
Inclusion Criteria:

* More than 3 months after stroke;
* Ischemic or hemorrhagic stroke with upper limb motor impairment;

Exclusion Criteria:

* Any contraindication for application of transcranial magnetic stimulation;
* Peripheral lesions in the assessed upper limb;
* Score ≤ 18 at Folstein Mini Mental State Examination;
* Alteration of drugs that alter the excitability of the cortex (in less than 3 months);
* Application of botulinum toxin in less than 6 months.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-03-29 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Brain symmetry (baseline) | Before each session (10 sessions for 5 days a week for two weeks)
  Accessed with:
  Quantitative electroencephalogram (qEEG) through the power spectral density (PSD) for each channel considering each band frequency: delta (0,5 a ≤ 4 Hz); theta (> 4 a ≤ 8 Hz); alpha (> 8 a ≤13 Hz); beta (> 13 a ≤ 30 Hz); gama (< 30 a ≤ 45 Hz) and the relative power for each band. . The Brain Symmetry Index (BSI) will be used to assess the absolute value of the difference in mean hemispheric power in the frequency range of 1 to 45Hz. All of these measures derive from each qEEG band frequency.
Brain symmetry (post-treatment) | After each session (10 sessions for 5 days a week for two weeks)
  Accessed with:
  Quantitative electroencephalogram (qEEG) through the power spectral density (PSD) for each channel considering each band frequency: delta (0,5 a ≤ 4 Hz); theta (> 4 a ≤ 8 Hz); alpha (> 8 a ≤13 Hz); beta (> 13 a ≤ 30 Hz); gama (< 30 a ≤ 45 Hz) and the relative power for each band. . The Brain Symmetry Index (BSI) will be used to assess the absolute value of the difference in mean hemispheric power in the frequency range of 1 to 45Hz. All of these measures derive from each qEEG band frequency.
Brain symmetry (baseline) | Before each session (10 sessions for 5 days a week for two weeks)
  Accessed with:
  Low-Resolution Brain Electromagnetic Tomography (LORETA) software. All data from qEEG will also be computed to the LORETA software to generate a tridimensional image of the patient's brain.
Brain symmetry (post-treatment) | After each session (10 sessions for 5 days a week for two weeks)
  Accessed with:
  Low-Resolution Brain Electromagnetic Tomography (LORETA) software. All data from qEEG will also be computed to the LORETA software to generate a tridimensional image of the patient's brain.

SECONDARY OUTCOMES:
Change in Fugl Meyer assesment of paretic upper limb motor function | 10 sessions (5 days a week for two weeks)
  Fugl Meyer assesment is used to measure motor control recovery. It is a 226 point scoring system that includes the following sessions: range of motion, pain, sensation,motor function of upper and lower limbs, balance, coordination and velocity. We will apply only two sessions: upper limb motor function and coordination/velocity, these sessions totalize 66 points. Higher scores indicates better outcomes
Modified Ashworth Scale | 10 sessions (5 days a week for two weeks)
  The modified Ashworth scale is a 6-point rating scale that is used to measure muscle tone and it will be used to determine the spasticity wrist flexor muscles in the affected hand by stroke. It evaluates the antagonist muscles that limits the force of agonist muscled during a intended motion.
The National Institutes of Health Stroke | 10 sessions (5 days a week for two weeks)
  This scale will determine the severity and disability level of the post-stroke patient; which consists of 15 items that assess the domains: level of consciousness, eye movements, visual field, facial movements, motor function and ataxia of upper and lower limbs, as well as sensitivity, language, presence of dysarthria and spatial neglect. Each domain punctuates a specific skill from 0 (zero) to 4 points that may vary until a maximum of 42 points.

CONTACTS AND LOCATIONS:
Locations (1):
- Federal University of Pernambucano, Recife, Pernambuco, Brazil